CLINICAL TRIAL: NCT04235725
Title: Implementation of Harmonized Depression Outcome Measures in a Primary Care Registry and a Mental Health Registry to Support Patient-Centered Outcomes Research
Brief Title: Implementation of Harmonized Depression Outcome Measures in a Primary Care Registry and a Mental Health Registry
Status: Completed | Type: Observational
Sponsor: OM1, Inc. (Industry)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AHRQ_DEP_Registry
Record Dates: First submitted 2020-01-07; First posted 2020-01-22 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Major Depression; Dysthymia
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Harmonized Depression Outcome Measures — This is an observational study where retrospective data on previous disease status and patient characteristics will be collected and combined with longitudinal data from these data sources on outcomes during the study timeframe.

SUMMARY:
The purpose of this pilot project is to demonstrate feasibility and value of collecting harmonized outcomes measures for major depressive disorder (MDD) in two registries and combining the data to support patient-centered outcomes research.

DETAILED DESCRIPTION:
The study is a longitudinal, multi-center observational feasibility study that will include data on eligible patients with a diagnosis of major depressive disorder (MDD). Retrospective data on previous disease status and patient characteristics will be collected and combined with longitudinal data from these data sources on outcomes during the study timeframe. All data will be collected from institution electronic medical records (EMRs), PRO portals, and other existing data sources, as needed.

Two registries (PsychPRO and the PRIME Registry) will participate in this feasibility study. A total of 20 sites participating in the registries (10 from each registry) will be recruited to participate in this study. To participate, sites must see adult patients with major depression or dysthymia and be willing to collect the PHQ-9 on a regular basis. Sites will have the option of using the Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER) scale to capture information on adverse events, but use of the FIBSER is not required.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Diagnosis of major depression or dysthymia as documented in the patient's EMR

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will collect data on approximately 200 patients with a diagnosis of major depression or dysthymia from a total of 20 sites (10 from each registry).
Sampling Method: Non-Probability Sample
Enrollment: 953 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Death from suicide | 12-month intervals
  Patient age 18 or older with a diagnosis of major depression or dysthymia who died from suicide.
Improvement in Depressive Symptoms: Remission | Baseline
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27.
Improvement in Depressive Symptoms: Remission | 6 months post baseline (+/- 60 days)
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27.
Improvement in Depressive Symptoms: Remission | 12 months post baseline (+/- 60 days)
  Patient Health Questionnaire-9 score > 9 who demonstrates remission defined as a Patient Health Questionnaire-9 score less than 5. Patient Health Questionnaire scores range from 0 to 27.
Improvement in Depressive Symptoms: Response | Baseline
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27.
Improvement in Depressive Symptoms: Response | 6 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27.
Improvement in Depressive Symptoms: Response | 12 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 score > 9 who demonstrates a response to treatment defined as a Patient Health Questionnaire-9 score that is reduced by 50% or greater from the initial Patient Health Questionnaire-9 score. Patient Health Questionnaire scores range from 0 to 27.
Worsening in Depressive Symptoms: Recurrence | Baseline
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27.
Worsening in Depressive Symptoms: Recurrence | 6 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27.
Worsening in Depressive Symptoms: Recurrence | 12 months post baseline (+/- 60 days)
  Patient age 18 or older with a diagnosis of major depression or dysthymia and an initial Patient Health Questionnaire-9 > 9 who demonstrates remission (defined as a Patient Health Questionnaire-9 score < 5) of at least two months' duration and subsequently experiences a recurrence of a depressive episode, defined as a Patient Health Questionnaire-9 score > 9 OR hospitalization for depression or suicidality. Patient Health Questionnaire scores range from 0 to 27.
Adverse Events | Baseline
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the EMR. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6.
Adverse Events | 6 months post baseline (+/- 60 days)
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the EMR. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6.
Adverse Events | 12 months post baseline (+/- 60 days)
  Depression treatment-related adverse events, captured using the Frequency, Intensity, and Burden of Side Effects Ratings scale where available and extracted from data routinely recorded in the EMR. The Frequency, Intensity, and Burden of Side Effects Ratings score ranges from 0 to 6.
Suicide Ideation and Behavior and Behavior | Baseline
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record.
Suicide Ideation and Behavior and Behavior | 6 months post baseline (+/- 60 days)
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record.
Suicide Ideation and Behavior and Behavior | 12 months post baseline (+/- 60 days)
  Selection of 'several days', 'more than half the days' or 'nearly every day' option on Patient Health Questionnaire-9 item 9 ("Thoughts that you would be better off dead or of hurting yourself in some way") and/or documentation of nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, or active suicidal ideation extracted from data routinely recorded in the Electronic Medical Record.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - American Psychiatric Association, Washington D.C., District of Columbia
  - American Board of Family Medicine, Lexington, Kentucky

REFERENCES:
- See also: AHRQ webpage containing details on this initiative — https://effectivehealthcare.ahrq.gov/products/registry-of-patient-registries/outcome-measure-harmonization